CLINICAL TRIAL: NCT05276167
Title: The Effect of Hyperthermic Intravesical Perfusion on the Risk of Intraoperative Implantation of Muscle-invasive Bladder Urothelial Carcinoma and Its Safety Analysis
Brief Title: Hyperthermic Intravesical Perfusion for Muscle-invasive Bladder Urothelial Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ytj20210926
Record Dates: First submitted 2021-11-24; First posted 2022-03-11 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-02

CONDITIONS: High-Risk, Non-Muscle Invasive Bladder Urothelial Carcinoma; Perfusion; Complications; Intraoperative Complications
MeSH Terms: conditions — Intraoperative Complications

STUDY DESIGN:
Intervention Model Description: The participants will be divided into two groups (the experimental group and control group). Participants in the experimental group will be treated with hyperthermic intravesical perfusion before receiving radical cystectomy. Participants in the control group will receive radical cystectomy alone.
Who Masked: Participant
Masking Description: The participants will be randomly (1:1) divided into the experimental and control groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental): Participants in the experimental group will be treated with hyperthermic intravesical perfusion before receiving radical cystectomy.
  Interventions: Device: hyperthermic intravesical perfusion
- The control group (No Intervention): Participants in the control group will receive radical cystectomy alone.

INTERVENTIONS:
Device: hyperthermic intravesical perfusion — Participants in the experimental group will be treated with hyperthermic intravesical perfusion before receiving radical cystectomy
  Arms: The experimental group

SUMMARY:
To evaluate the effect of hyperthermic intravesical perfusion on the risk of intraoperative implantation of muscle-invasive bladder urothelial carcinoma and its safety.

DETAILED DESCRIPTION:
The participants will be divided into two groups (the experimental group and control group). Participants in the experimental group will be treated with hyperthermic intravesical perfusion before receiving radical cystectomy. Participants in the control group will receive radical cystectomy alone.

After follow-up, the effect of hyperthermic intravesical perfusion on the risk of intraoperative implantation of muscle-invasive bladder urothelial carcinoma and its safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* 18-75 years of age on day of signing informed consent.
* Have histologically confirmed muscle invasive disease of the urinary bladder.
* Histology must be urothelial carcinoma (transitional cell carcinoma) or urothelial carcinoma with mixed histology/features.
* Clinical stage II-III and Have a surgical evaluation that documents the plan for multimodality therapy with a consolidative radical cystectomy.
* Eastern Cooperative Oncology Group 0-1 and good organ function.

Exclusion Criteria:

* A non-surgical approach recommended by the treating urologist due to any reason.
* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 28 days prior to study registration.
* Has a diagnosis of immunodeficiency or received systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to study registration.
* Has a known additional malignancy that is progressing or required treatment ≤ 48 months of study registration. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has an active autoimmune disease requiring systemic treatment.
* Has known evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-programmed cell death 1, anti-programmed cell death-Ligand 1 antibody.
* Has a known history of Human Immunodeficiency Virus.
* Has known active Hepatitis B or Hepatitis C.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of intraoperative tumor cell dissemination | 3 years
  The rate of intraoperative tumor cell dissemination will be evaluated by lavage cytology of operating field

SECONDARY OUTCOMES:
Time to disease progression | 3 years
  Disease progression was defined as recurrence or metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- BR-PRG, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No